CLINICAL TRIAL: NCT03788603
Title: An Open Label, Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Rogaratinib (BAY1163877) in Chinese Patients With FGFR-positive Refractory, Locally Advanced, or Metastatic Solid Tumors
Brief Title: Rogaratinib (BAY1163877) in Chinese Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19177
Record Dates: First submitted 2018-12-19; First posted 2018-12-27 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Rogaratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rogaratinib (BAY1163877) (Experimental): Eligible patients will be selected based on the confirmation of high fibroblast growth factor receptor (FGFR) 1, 2, 3 or 4 mRNA expression levels in archival or fresh tumor biopsy specimens collected before the start of screening
  Interventions: Drug: Rogaratinib (BAY1163877)

INTERVENTIONS:
Drug: Rogaratinib (BAY1163877) — Rogaratinib will be administered on 20 days in Cycle 1 (single dosing on Day 1 and twice daily dosing on Days 3-21). In Cycles ≥2, rogaratinib will be administered twice daily for 21 days, with cycles repeated every 21 days. Treatment will be continued until death, tumor progression, unacceptable toxicity, consent withdrawal, or until another criterion is met for withdrawal from the study at the discretion of the investigator.

SUMMARY:
This study is planned to determine the safety and tolerability of rogaratinib in Chinese patients with fibroblast growth factor receptor (FGFR)-positive refractory, locally advanced, or metastatic solid tumors and to characterize the pharmacokinetics of rogaratinib in Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years of age on the date of signing the Main Informed Consent Form.
* Subjects with histologically or cytologically confirmed, refractory, locally advanced, or metastatic solid tumors who are not candidates for any standard therapy, excluding primary brain or spinal tumors.
* High FGFR1, 2, 3 or 4 mRNA expression levels based on archival or fresh tumor biopsy specimen analysis (RNAscope score of 3 or 4)
* At least one measurable lesion outside the central nervous system according to Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1) A lesion in a previously irradiated area is eligible and to be considered measurable disease as long as there is objective evidence of progression of the lesion prior to study enrollment. Patients with resected primary tumors who have documented metastases are eligible.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 or 1
* Life expectancy of at least 3 months
* Adequate bone marrow, liver and renal function as assessed by laboratory requirements conducted within 7 days before the first dose of rogaratinib:

  * Hemoglobin (Hb) ≥9.0 g/dL (without transfusion or erythropoietin within 4 weeks before screening)
  * Absolute neutrophil count (ANC) ≥1,500/mm3
  * Platelet count ≥100,000/mm3
  * Total bilirubin ≤1.5 times the upper limit of normal (ULN). Documented or diagnosed constitutional jaundice such as Gilbert syndrome is allowed if total bilirubin is mildly elevated (<6 mg/dL).
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times ULN (≤5 times ULN for patients with liver involvement of their cancer)
  * Alkaline phosphatase ≤2.5 times ULN (≤5 times ULN for patients with liver involvement of their cancer)
  * Amylase and lipase ≤2.5 times ULN
  * Serum creatinine ≤1.5 x ULN and glomerular filtration rate (GFR) ≥30 mL/min/1.73 m2, according to the Modified Diet in Renal Disease (MDRD) abbreviated formula

Exclusion Criteria:

- Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study.

The following previous or concurrent cancer types might be acceptable: cervical carcinoma in situ, treated basal cell carcinoma, locally confined prostate cancer, or any cancer curatively treated >3 years before the start of rogaratinib.

- Symptomatic brain or meningeal or spinal metastases.

Asymptomatic brain or meningeal or spinal metastases are acceptable if all of the following criteria are met:

* Definitive therapy completed >6 months before the start of rogaratinib
* No evidence of the growth of brain or meningeal or spinal metastases on an imaging test performed within 4 weeks before the start of rogaratinib
* Clinically and radiologically stable with respect to the tumor at the time of study entry

  * Moderate or severe liver cirrhosis (Child-Pugh class B or C)
  * History or current evidence of altered endocrine regulation of calcium phosphate homeostasis (e.g. parathyroidectomy, parathyroid disorder, tumor lysis, tumoral calcinosis)
  * Any previous drug / procedure-related toxicity (patients with persistent alopecia, anemia, and / or hypothyroidism can be included) not recovered to National Cancer Institute's Common Terminology Criteria for Adverse Event, version 4.03 (CTCAE v4.03) Grade 0 or 1 or not recovered to baseline preceding the prior treatment
  * Current diagnosis of any retinal disorders including retinal detachment, retinal pigment epithelial detachment (RPED), serous retinopathy or retinal vein occlusion.
  * Previous treatment with anti-FGFR directed therapies (e.g. receptor tyrosine kinase inhibitors including rogaratinib or FGFR-specific antibodies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-04-14 (Actual)

PRIMARY OUTCOMES:
Frequency of Treatment-Emergent Adverse Events(TEAEs) | 30 days after last dose of rogaratinib
Severity of Treatment-Emergent Adverse Events(TEAEs) | 30 days after last dose of rogaratinib
Cmax: Maximum drug concentration in plasma after dose administration | Cycle 1 Day 1 (each cycle is 21 days)
  Single dose
AUC(0-12): AUC from time zero to 12 hours p.a. after first-dose administration | Cycle 1 Day 1 (each cycle is 21 days)
  Single dose
Cmax,md: Cmax after multiple dosing | Cycle 1 Day 15 (each cycle is 21 days)
  Multiple dose
AUC(0-12)md: AUC(0-12) after multiple dosing | Cycle 1 Day 15 (each cycle is 21 days)
  Multiple dose

SECONDARY OUTCOMES:
Phosphate levels | Within 7-14 days after the last dose of rogaratinib
Response rate | Within 7-14 days after the last dose of rogaratinib
  Response rate is defined as the proportion of patients who have a best overall response rating of complete response (CR) and partial response (PR) that is achieved during treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/